CLINICAL TRIAL: NCT03668145
Title: Mesenchymal Stem Cell Transplantation for Refractory Primary Biliary Cholangitis, a Randomized Double-blind Placebo Controlled Trial
Brief Title: Mesenchymal Stem Cell Transplantation for Refractory Primary Biliary Cholangitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Prof. Dr., Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20172050-1
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis (now termed as primary biliary cholangitis), mesenchymal stem cell,
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be blinded to participant, care provider, investigator and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC group (Experimental): mesenchymal stem cell transplantation via peripheral vein: 0.1-1x10E6 MSCs/kg body weight administered via peripheral vein at week 0, 4, 8 plus UDCA.
  Interventions: Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein
- control (Placebo Comparator): placebo infusions (placebo infusion differs from the experimental infusion in only that placebo has no mesenchymal stem cells) will be administered via peripheral vein at week 0, 4, 8 plus UDCA.
  Interventions: Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein

INTERVENTIONS:
Procedure: mesenchymal stem cell transplantation or placebo infusion via peripheral vein — 0.1-1x10E6 MSCs/kg body weight will be administered via peripheral vein for 3 times at week 0, 4 and 8 mesenchymal stem cell mesenchymal stem cell infusion produced by Cell products of National Engineering Research Center(short for CPNERC), Tianjin, China For control group, placebo infusions will be given to the participants at the same time points

SUMMARY:
Ursodeoxycholic acid is the mainstay treatment medicine for primary biliary cholangitis(PBC). About 1/3 of the patients do not respond to UDCA, which is defined as refractory PBC. Mesenchymal stem cells (MSC) has been reported to improve the outcomes of PBC patients. Randomization controlled studies are needed to confirm the long term effect of MSC treatment for refractory PBC. This study aimed to investigate the safety and efficacy of mesenchymal stem cells in PBC patients that do not respond to UDCA treatment. This study is an double-blind multicenter randomized and placebo-controlled study. Patients with with refractory PBC will be randomly assigned to receive MSC treatment plus UDCA or UDCA alone (control). Three times of MSC infusion (0.1-1x10E6 cells/kg body weight) via peripheral vein will be given to the experimental group (once in 4 weeks). The primary outcome is absolute change in alkaline phosphatase. Secondary outcomes are changes of other liver function indices such as ALT TBIL AST GGT, improve of symptoms and liver histology.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. Age between 18-70 years old
3. BMI between 17-28
4. Meeting at least 2 of the 3 criteria: (1) positive for anti-mitochondial antibody (AMA)；(2) Elevated ALP or GGT；(3) PBC diagnosis confirmed by liver biopsy
5. Serum ALP >/=1.67 ULN after at leat 6 months treatment with UDCA 1(3-17mg/kg/day) -

Exclusion Criteria:

1. Pregnancy, breast-feeding females
2. Use of liver-toxic drugs over 2 week within 6 months prior to recruitment；
3. refractory variceal bleeding, uncontrolled hepatoencephalopathy or uncontrolled ascites.
4. Acute of chronic kidney failure.
5. Commodities with other liver diseases such as viral hepatitis, alcoholic liver disease, auto-immune hepatitis or liver cancer
6. Severe cardiovascular disease；
7. liver transplantation listed patients；
8. ALT/AST over 5xULN，or total bilirubin >85umol/l
9. anticipated need for liver transplantation within 1 year according to mayo risk score
10. Other candidates who are judged to be not applicable to this study by doctors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of alkaline phosphatase (ALP) | 1 year
  The absolute value change of ALP after 1 year of the initial stem cell treatment

SECONDARY OUTCOMES:
Change of other liver function indices | 1 year
  The absolute value change of total bilirubin, ALT, AST, GGT after initial stem cell treatment
Change of liver histology | 1 year
  histological scores assessed by liver biopsy at baseline and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Changcun Guo, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: The data will be available after the completion of the study and before publications for 1 year